CLINICAL TRIAL: NCT05017389
Title: A Cohort Study on the Long-term Health Outcomes of Premature Infants
Brief Title: Long Term Health Cohort of Premature Infants
Status: Recruiting | Type: Observational
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Principal Investigator, BeiFei, director of neonatology department, Shanghai Children's Medical Center
Other Study IDs: LY-SCMC2020-01
Record Dates: First submitted 2021-07-27; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Take 2-5ml blood samples for relevant biochemical tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Griffiths development scales — Griffiths development scales Chinese Edition (gds-c) was used to evaluate the development levels of children up to 6 years and WISC for children more than 6 years.
  Other Names: Wechsler Intelligence Scale

SUMMARY:
Establish a clinical diagnosis and treatment and long-term follow-up database of preterm infants, and analyze the effects of prenatal factors (including genetic characteristics, maternal diseases, etc.), postnatal diagnosis and treatment measures and family maintenance environment after discharge on preterm infant mortality and major diseases in the near and long term.

DETAILED DESCRIPTION:
As an increasing large group, the long-term quality of life and health status of preterm infants have become a very important public health problem in China. This cohort study is a single center clinical cohort study. By collecting the clinical diagnosis, treatment and follow-up data of preterm infants admitted to the neonatal department of our hospital for 3 consecutive years (about 1200 cases), and following them for 18 years, a relatively complete resource database for the long-term health and development of preterm infants is established. The effects of perinatal factors, diagnosis and treatment methods and family rearing environment on the survival rate, neurointelligence development, chronic metabolic diseases and respiratory diseases of preterm infants were analyzed. It provides a basis for further improving the diagnosis and treatment plan, exploring potential therapeutic targets and establishing prediction models.

ELIGIBILITY:
Inclusion Criteria:

1. Live born newborns with gestational age ≤ 36 + 6 weeks
2. Transfer to the neonatal ward of Shanghai Children's medical center within 24 hours after birth
3. Those who have lived in Shanghai for more than 1 year and plan to live in Shanghai for a long time. Parents voluntarily participated in the study and signed informed consent

Exclusion Criteria:

1. Premature infants: termination of treatment due to family factors (non-disease reasons) and hospitalization time ≤ 2 weeks
2. Major congenital malformations
3. Parents refuse to participate in the study

Ages: 15 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: premature infants with gestational age ≤ 36 + 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
neural development at 1 year old | 1 year
  Taking Griffiths development scales Chinese Edition test for all the participants.
neural development at 2 years old | 2 years
  Taking Griffiths development scales Chinese Edition test for partial participants.
neural development at 6 years old | 6 years
  Taking Wechsler Intelligence Scale for participants.
Growth and neural development at 12 years old | 12 years
  Taking Wechsler Intelligence Scale for participants.
Growth and neural development at 18 years old | 18 years
  Taking Wechsler Intelligence Scale for participants.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Bei, Ph.D, Study Chair — Shanghai Children's Medical Center
Locations (1):
- Shanghai children's medical center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No